CLINICAL TRIAL: NCT04725981
Title: Vaginal Stump Infection After Total Laparoscopic or Robot-assisted Hysterectomy
Brief Title: Vaginal Stump Infection After Laparoscopic Hysterectomy
Acronym: CoToIn
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Spital Limmattal Schlieren (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Tatiana Naydina Ragaz, Senior Gynecologist in Women's Clinic, Spital Limmattal Schlieren
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-Nr.2018-00777
Record Dates: First submitted 2020-12-08; First posted 2021-01-27 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Laparoscopic Hysterectomy; Vaginal Infection
Keywords: vaginal closure technique
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Intervention Model Description: Compare two surgical techniques Prospective randomized, controlled, single-blind inversion study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (test surgical technique) (Experimental): Colpotomy closure technique: 3 Z-suture with PDS 0 and 1 continuous suture with V-Loc 2-0
  Interventions: Procedure: Total laparoscopic hysterectomy
- Arm B (control surgical technique) (Active Comparator): Colpotomy closure technique: 3 Z-suture with PDS 0
  Interventions: Procedure: Total laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Total laparoscopic hysterectomy — Control group: colpotomy closure technique: 3 Z-sutures PDS 0 Intervention group: colpotomy closure technique: 3 Z sutures with PDS 0 and 1 continuous suture with V-Loc 2-0

SUMMARY:
Comparing two surgical techniques in relation to vaginal stump infection, analysis of patient-based and therapy-based risk factors.

DETAILED DESCRIPTION:
Comparing two surgical techniques for vaginal stump infection after total laparoscopic or robot-assisted hysterectomy. Analysis of patient-based and therapy-based risk factors with the aim of optimizing the surgical technique and objectifying the risk factors. Control group: old colpotomy technique (3 Z-sutures PDS 0); Intervention group: new colpotomy technique (3 Z sutures with PDS 0 and 1 continuous suture with V-Loc 2-0)

ELIGIBILITY:
Inclusion Criteria:

1. Patient > = 18 years old
2. Indication for total laparoscopic or robot-assisted hysterectomy
3. Benign uterine disease
4. Signed informed consent for study participation

Exclusion Criteria:

1. Patient with malignant gynecological diseases
2. Combination with other abdominal / vaginal interventions, except:

   * Adhesiolysis
   * Endometriosis removal (without rectovaginal endometriosis)
   * Conization
   * Hysteroscopy / curettage
3. Immunosuppressive therapy with cytostatics, glucocorticoids, HIV
4. Bleeding tendency / haemophilia
5. Acute infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All patients> 18 years of age with an indication for total laparoscopic or robot-assisted hysterectomy (with or without adnexa / tubes) for benign uterine diseases.
Enrollment: 141 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with vaginal stump infection in intervention group and control group | 6 weeks
  7.-10. day and 6 weeks postoperatively:
  1. T ° C (fever> = 38 ° C)
  2. blood pressure (mm Hg)
  3. general condition (good, reduced, bad)
  4. Speculum examination / condition of the colpotomy:
     * non-irritating / intact
     * dehiscent
     * bleeding
     * fibrin-coated
     * purulent
     * tender
     * hyperemic
     * Infiltrated
     * Fistula formation
  5. Lower abdominal pain (Visual Analog Scale (VAS): 0-10
  6. transvaginal sonography: encapsulated RF on vaginal stump J: ☐N: ☐
  7. Laboratory CRP (> 10mg / L) Hb (<120 g / L) Lc ( >10 G / L)
  The diagnosis of vaginal stump infection was made based on 2 of 3 positive clinical symptoms, 1 additional criterion and the corresponding sonographic findings.
  I. Clinical symptoms: 1. Fever> = 38 ° C; 2. Dolence, redness, swelling, pus in the colpotomy area; 3. Lower abdominal pain ( VAS >5) II. Sonographic signs (TVUS): encapsulated cystic mass on the vaginal stump Additional criteria: 1. CRP increased (> 10mg / l); 2. Antibiotic therapy needs

SECONDARY OUTCOMES:
Identify of patient-based and treatment-based risk factors for vaginal stump infection. | 6 weeks
  connection between Obesity ( BMI >30 kg/ m2), nicotine abuse ( >5 cigarettes/d), anemia ( Hb <120g/L), operation time ( >120min), uterine volume ( >100 cm3) and appearance of vaginal stump infection

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Naydina Ragaz, Principal Investigator — Tatiana Naydina Ragaz, Deputy Senior Gynecologist Women's Clinic, Spital Limmattal, Zurich Schlieren
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No